CLINICAL TRIAL: NCT01987505
Title: Open Label, Single-arm, Phase IIIb Clinical Trial to Evaluate the Safety of Switching From Intravenous Rituximab to Subcutaneous Rituximab During First Line Treatment for CD20+ Non-Hodgkin's Follicular Lymphoma and Diffuse Large B-cell Lymphoma.
Brief Title: MabRella Study: A Study to Evaluate the Safety of Switching From Intravenous to Subcutaneous Administration of Rituximab During First-Line Treatment for Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28943; 2013-001118-14 (EudraCT Number)
Record Dates: First submitted 2013-11-08; First posted 2013-11-19 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Lymphoma, Non Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Subcutaneous Rituximab (Experimental): Participants with CD20+ non-Hodgkin's follicular lymphoma (FL) or diffuse large B-cell lymphoma (DLBCL), who had already received at least one full dose of intravenous (IV) rituximab will be treated with subcutaneous (SC) rituximab. Participants with FL will be administered 1400 mg rituximab during induction therapy (once monthly for 4-7 cycles) and maintenance therapy (once every 2 months for 6-12 cycles). Participants with DLBCL will be administered 1400 mg SC of rituximab once monthly for 4-7 cycles. Treatment duration is expected to last up to 7 months for participants with DLBCL and up to 32 months for participants with FL.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 1400 mg will be injected subcutaneously (SC).
  Other Names: MabThera; Rituxan

SUMMARY:
This open-label, single-arm, phase IIIb study will evaluate the safety of switching from intravenous (IV) to subcutaneous (SC) administration of rituximab during first-line treatment for participants with CD20+ non-Hodgkin's follicular lymphoma (FL) or diffuse large B-cell lymphoma (DLBCL) who have already received at least one full dose of rituximab IV. Participants with FL will be given 1400 mg rituximab SC during induction therapy (once monthly for 4-7 cycles) and maintenance therapy (once every 2 months for 6-12 cycles). 1400 mg SC of rituximab will be given to participants with DLBCL once monthly for 4-7 cycles. Treatment duration is expected to last up to 7 months for participants with DLBCL and up to 32 months for participants with FL.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years at time of enrolment.
* Life expectancy ≥ 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3.
* Fertile men or women of childbearing potential must use effective contraception until at least 12 months after the last dose; women must not be pregnant.
* Histologically confirmed CD20+ diffuse large B-cell lymphoma (DLBCL) or CD20+ follicular Non-Hodgkin Lymphoma (FL) grade 1, 2 or 3a according to the World Health Organisation Classification system.

Induction only:

* Participants with Follicular Lymphoma should meet Groupe D'Etude des Lymphomes Folliculaires (GELF) criteria to initiate treatment.
* At least tumor >/= 1.5 cm as measured by computed tomography (CT) scan.

FL treatment-related criteria

- Currently being treated with rituximab IV during first-line therapy and has received at least one full dose of rituximab IV.

Exclusion Criteria:

* Transformed lymphoma.
* Primary central nervous system lymphoma, primary effusion lymphoma, primary mediastinal DLBCL, DLBCL of the testis, primary cutaneous DLBCL or histologic evidence of transformation to a Burkitt lymphoma.
* History of other cancer, including one that has been treated but not with curative intent, unless the cancer has been in remission without treatment for >/= 5 years prior to dosing. Note: Participants with a history of cured skin cancer or in situ carcinoma of the cervix are eligible for the study.
* Ongoing corticosteroid use > 30 mg/day of prednisone or equivalent. Note: Participants receiving corticosteroid treatment with </= 30 mg/day of prednisone or equivalent must be on a stable regimen for at least 4 weeks prior to start of dosing.
* Inadequate renal, hematologic, or hepatic function.
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products.
* For participants with DLBCL: Contraindication to any of the individual components of CHOP (cyclophosphamide, vincristine, doxorubicin and prednisone), including prior anthracycline treatment.
* For participants with FL: contraindication to standard chemotherapy.
* Other serious underlying medical conditions.
* Recent major surgery (within 4 weeks prior to dosing), other than for diagnosis.
* Active and/or severe infections (excluding nail fungal infections) or any infection requiring treatment with IV antibiotics or hospitalization within 4 weeks prior to dosing.
* Active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection. Note: Participants testing positive for Hepatitis B or C virus antibodies but with an undetectable viral load may be included.
* History of Human Immunodeficiency Virus (HIV) positive status.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- Spain (39):
  - Hospital De Txagorritxu; Servicio de Hematologia, Vitoria-Gasteiz, Alava
  - Hospital General de Elda; Servicio de Hematologia, Elda, Alicante
  - Hospital Son Llatzer; Servicio de Hematologia, Palma de Mallorca, Balearic Islands
  - Hospital de Granollers, Servicio de Hematología, Granollers, Barcelona
  - Hospital Mutua de Terrassa; Servicio de Hematologia, Terrassa, Barcelona
  - Hospital General de Castellon; Servicio de Hematologia, Castellon, Castellon
  - Complejo Hospitalario Universitario A Coruña (CHUAC); Servicio de Hematologia, A Coruña, LA Coruña
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Hematologia, Santiago de Compostela, LA Coruña
  - Complejo Hospitalario San Millan - San Pedro; Servicio Hematologia, Logroño, La Rioja
  - Complejo Asistencial de León, Servicio de Hematología, León, LEON
  - Hospital Universitario de Fuenlabrada; Servicio de Hematologia, Fuenlabrada, Madrid
  - Hospital Severo Ochoa; Servicio de Hematologia, Leganés, Madrid
  - Hosital Universitario de Mostoles;Servicio de Hematologia, Móstoles, Madrid
  - Clinica Universitaria de Navarra; Servicio de Hematologia, Pamplona, Navarre
  - Hospital de Navarra, Servicio de Hematología, Pamplona, Navarre
  - Complejo Hospitalario Universitario de Vigo; Servicio de Hematologia, Vigo, Pontevedra
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Oncologia, Santa Cruz de Tenerife, Tenerife
  - Hospital de Basurto; Servicio de Hematologia, Bilbao, Vizcaya
  - Hospital de Galdakano; Servicio de Hematologia, Galdakao, Vizcaya
  - Complejo Hospitalario Torrecardenas; Servicio de Hematologia, Almería
  - Hospital Universitario de Burgos, Servicio de Hematología, Burgos
  - Hospital Universitario Reina Sofia; Servicio de Hematologia, Córdoba
  - Hospital Universitario Virgen de las Nieves; Servicio de Hematologia, Granada
  - Hospital Universitario de Gaudalajara; Hematología, Guadalajara
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Hematologia, Lleida
  - Hospital Infanta Leonor; Servicio de Hematologia, Madrid
  - Fundacion Jimenez Diaz; Servicio de Hematologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Hematología, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio Hematologia, Madrid
  - Hospital Universitario Puerta de Hierro; Servicio de Hematologia, Madrid
  - Hospital Universitario Principe de Asturias; Servicio de Hematología, Madrid
  - Hospital Univ. Virgen de la Victoria, Málaga
  - Hospital General Universitario J.M Morales Meseguer; Servicio de Hematología, Murcia
  - Hospital Universitario Virgen de Arrixaca; Servicio de Hematologia, Murcia
  - Complejo Hospitalario de Pontevedra; Servicio de Hematologia, Pontevedra
  - Complejo Asistencial de Segovia, Segovia
  - Hospital Universitario Virgen Macarena; Servicio de Hematologia, Seville
  - Hospital Univ. Nuestra Señora de Valme; Servicio de Hematologia, Seville
  - Hospital de Rio Hortega; Servicio de Hematologia, Valladolid

REFERENCES:
- [Derived] Petrini M, Gaidano G, Mengarelli A, Consoli U, Santoro A, Liberati AM, Ladetto M, Fraticelli V, Guarini A, Mannina D, Ferrando P, Corradini P, Musto P, Stelitano C, Marino D, Camera A, Murineddu M, Battistini R, Caparrotti G, Turrini M, Arcaini L, Santini S, Cerqueti M, Ferreri AJM, Cantore N, Inzoli A, Cardinale G, Ronci B, La Nasa G, Massimi S, Gaglione G, Barbiero V, Martelli M. Safety and Efficacy of Subcutaneous Rituximab in Previously Untreated Patients with CD20+ Diffuse Large B-Cell Lymphoma or Follicular Lymphoma: Results from an Italian Phase IIIb Study. Adv Hematol. 2022 Jan 27;2022:5581772. doi: 10.1155/2022/5581772. eCollection 2022. PMID 35126524
- [Derived] Garcia-Munoz R, Quero C, Perez-Persona E, Domingo-Garcia A, Perez-Lopez C, Villaescusa-de-la-Rosa T, Martinez-Castro AM, Arguinano-Perez JM, Parra-Cuadrado JF, Panizo C. Safety of switching from intravenous to subcutaneous rituximab during first-line treatment of patients with non-Hodgkin lymphoma: the Spanish population of the MabRella study. Br J Haematol. 2020 Mar;188(5):661-673. doi: 10.1111/bjh.16227. Epub 2019 Oct 1. PMID 31573078

RESULTS

PARTICIPANT FLOW:
Groups:
- Subcutaneous Rituximab: Participants with CD20+ non-Hodgkin's follicular lymphoma (FL) or diffuse large B-cell lymphoma (DLBCL), who had already received at least one full dose of intravenous (IV) rituximab were treated with subcutaneous (SC) rituximab during first-line treatment. Participants with FL were administered 1400 mg rituximab during induction therapy (once monthly for 4-7 cycles) and maintenance therapy (once every 2 months for 6-12 cycles). Participants with DLBCL were administered 1400 mg SC of rituximab once monthly for 4-7 cycles. Treatment duration was expected to last up to 7 months for participants with DLBCL and up to 32 months for participants with FL.
Period: Overall Study
Arm/Group | Subcutaneous Rituximab
Started | 140
Completed | 106
Not Completed | 34
Not completed — Other | 9
Not completed — Withdrawal by Subject | 2
Not completed — Other Reason | 2
Not completed — Lost to Follow-up | 15
Not completed — Investigator Decision | 2
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all enrolled participants. All analyses described have been performed by type of lymphoma (DLBCL/ FL) and overall.
Groups:
- Diffuse Large B-Cell Lymphoma: Participants with diffuse large B-cell lymphoma (DLBCL), who had already received at least one full dose of intravenous (IV) rituximab were treated with subcutaneous (SC) rituximab. Participants with DLBCL were administered 1400 mg SC of rituximab once monthly for 4-7 cycles. Treatment duration was expected to last up to 7 months for participants with DLBCL.
- Follicular Lymphoma: Participants with CD20+ non-Hodgkin's follicular lymphoma (FL), who had already received at least one full dose of intravenous (IV) rituximab were treated with subcutaneous (SC) rituximab. Participants with FL were administered 1400 mg rituximab during induction therapy (once monthly for 4-7 cycles) and maintenance therapy (once every 2 months for 6-12 cycles). Treatment duration was expected to last to 32 months for participants with FL.
- Total: Total of all reporting groups
Arm/Group | Diffuse Large B-Cell Lymphoma | Follicular Lymphoma | Total
Number analyzed (Participants) | 29 | 111 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (12.0) | 59.6 (12.5) | 60.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 58 | 75
  Male | 12 | 53 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 0 | 1 | 1
  Caucasian | 29 | 110 | 139

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Administration-Associated Reactions (AARs)
Description: AARs were defined as all adverse events (AEs) occurring within 24 hours of rituximab SC administration and which were considered related to study drug. AARs included infusion/injection-related reactions (IIRRs), injection-site reactions, administration site conditions and all symptoms thereof. Grading was completed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
Time Frame: From start of treatment to end of treatment (up to 32 months)
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Groups:
- Diffuse Large B-Cell Lymphoma (DLBCL): Participants with diffuse large B-cell lymphoma (DLBCL), who had already received at least one full dose of intravenous (IV) rituximab were treated with subcutaneous (SC) rituximab. Participants with DLBCL were administered 1400 mg SC of rituximab once monthly for 4-7 cycles. Treatment duration was expected to last up to 7 months for participants with DLBCL.
- Follicular Lymphoma (FL): Participants with CD20+ non-Hodgkin's follicular lymphoma (FL), who had already received at least one full dose of intravenous (IV) rituximab were treated with subcutaneous (SC) rituximab. Participants with FL were administered 1400 mg rituximab during induction therapy (once monthly for 4-7 cycles) and maintenance therapy (once every 2 months for 6-12 cycles). Treatment duration was expected to last to 32 months for participants with FL.
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous Rituximab
Number analyzed (Participants) | 29 | 111 | 140
percentage of participants
  At Least One AAR | 34.5 | 52.3 | 48.6
  At Least One AAR Grade ≥ 3 | 0 | 2.7 | 2.1
  At Least One Serious AARs | 0 | 1.8 | 1.4
  Generalised or Remote from the Injection Site AARs | 57.9 | 11.1 | 15.1
  Localised at the injection site AARs | 42.1 | 88.9 | 84.9

2. Secondary Outcome: Percentage of Participants With At Least One Grade >/= 3 Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsen during a study are also considered as adverse events. Grading was completed according to the CTCAE, version 4.0.
Time Frame: From start of recruitment (10 months period) up to end of treatment at 32 months (total period up to 42 months)
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous Rituximab
Number analyzed (Participants) | 29 | 111 | 140
percentage of participants | 48.3 | 36.0 | 38.6

3. Secondary Outcome: Percentage of Participants With At Least One Grade >/= 3 Infusion/ Injection Related Reactions (IIRRs)
Description: Grading of IIRRs was completed according to the CTCAE, version 4.0.
Time Frame: From start of treatment to end of treatment (up to 32 months)
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous Rituximab
Number analyzed (Participants) | 29 | 111 | 140
percentage of participants | 0.0 | 2.7 | 2.1

4. Secondary Outcome: Percentage of Participants With At Least One Serious Adverse Event (SAE)
Description: SAE was defined as any experience that suggested a significant hazard, contraindication, side effect, or precaution, and fulfilled any of the following criteria: fatal (resulted in death), life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/ birth defect, was medically significant or required intervention to prevent any of the other outcomes listed here.
Time Frame: From start of recruitment (10 months period) up to end of treatment at 32 months (total period up to 42 months)
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous Rituximab
Number analyzed (Participants) | 29 | 111 | 140
percentage of participants | 37.9 | 27.9 | 30.0

5. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the time from first dose of rituximab IV to first occurrence of progressive disease (PD) or relapse, according to the International Working Group (IWG) response criteria or initiation of a non-protocol-specified anti-lymphoma therapy or death, whichever occurs first. PD: >/= 50% increase lymph nodes and nodal mass size, any new lesion, enlarged liver/spleen, reappearance bone marrow abnormalities.
Time Frame: From time of first dose of rituximab IV before study enrollment up to end of study (up to approximately 62 months)
Population: Intent-to-Treat (ITT) population included all enrolled participants.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous Rituximab
Number analyzed (Participants) | 29 | 111 | 140
months | 25.79 [20.800 to 30.776] | 54.39 [51.416 to 57.362] | 52.314 [49.162 to 55.466]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from first dose of rituximab IV to the first occurrence of progressive disease (PD) or relapse, according to the International Working Group (IWG) response criteria or death from any cause. PD: >/= 50% increase lymph nodes and nodal mass size, any new lesion, enlarged liver/spleen, reappearance bone marrow abnormalities.
Time Frame: From time of first dose of rituximab IV before study enrollment up to end of study (up to approximately 62 months)
Population: ITT population included all enrolled participants.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous Rituximab
Number analyzed (Participants) | 29 | 111 | 140
months | 27.952 [23.443 to 32.460] | 54.389 [51.416 to 57.362] | 53.118 [50.108 to 56.127]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of rituximab IV to death from any cause.
Time Frame: From time of first dose of rituximab IV before study enrollment up to end of study (up to approximately 62 months)
Population: ITT population included all enrolled participants.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous Rituximab
Number analyzed (Participants) | 29 | 111 | 140
months | 37.42 [33.354 to 41.485] | 60.61 [59.692 to 61.535] | 59.516 [57.999 to 61.033]

8. Secondary Outcome: Disease-Free Survival (DFS)
Description: DFS was assessed in participants achieving complete response (CR) including complete response unconfirmed (Cru) and was defined as the period from the date of the initial CR/CRu until the date of relapse or death from any cause. CR: 1) disappearance of all evidence/symptoms of disease, 2) lymph nodes and nodal masses normal size, 3) enlarged spleen must have regressed in size, 4) normal bone marrow; CRu: see 1) and 3) of CR plus > 75% decrease in residual lymph node mass, indeterminate bone marrow. Reported here is the truncated mean estimate based on Kaplan-Meier analysis.
Time Frame: From time of first dose of rituximab IV before study enrollment up to end of study (up to approximately 62 months)
Population: ITT population included all enrolled participants.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous Rituximab
Number analyzed (Participants) | 29 | 111 | 140
months | 26.062 [23.510 to 28.613] | NA [NA to NA] — No events in this arm, therefore mean and 95% Confidence Interval could not be calculated. | 33.044 [31.489 to 34.600]

9. Secondary Outcome: Treatment Response Rate
Description: Treatment response rate was classified according to the International Working Group (IWG) response criteria: CR/Cru, partial response (PR), stable disease (SD) and PD. CR: 1) disappearance of all evidence/symptoms of disease, 2) lymph nodes and nodal masses normal size, 3) enlarged spleen must have regressed in size, 4) normal bone marrow; CRu: see 1) and 3) of CR plus > 75% decrease in residual lymph node mass, indeterminate bone marrow; PR: >/= 50% decrease lymph nodes and nodal mass size; decrease in liver/spleen size, no new sites; SD: less than a PR, but is not PD; PD: >/= 50% increase lymph nodes and nodal mass size, any new lesion, enlarged liver/spleen, reappearance bone marrow abnormalities.
Time Frame: 4-6 weeks after the last dose of Induction (Up to approximately 8 months)
Population: ITT population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous Rituximab
Number analyzed (Participants) | 29 | 111 | 140
percentage of participants
  Complete Response (CR) | 62.1 | 66.7 | 64.3
  Complete Response Unconfirmed (CRU) | 3.4 | 7.4 | 5.4
  Partial Response (PR) | 3.4 | 11.1 | 7.1
  Stable Disease (SD) | 0.0 | 3.7 | 1.8
  Progressive disease (PD) | 17.2 | 7.4 | 12.5
  Unable to Assess (UA) | 6.9 | 0.0 | 3.6
  Not Evaluable | 6.9 | 3.7 | 5.4

ADVERSE EVENTS:
Time Frame: From start of recruitment (10 months period) up to end of treatment at 32 months (total period up to 42 months)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. Safety Population included all enrolled participants who received at least one dose of study medication.
Arm/Group | Subcutaneous Rituximab
All-Cause Mortality (participants affected / at risk) | 4/140
Serious Adverse Events (participants affected / at risk) | 42/140
Other Adverse Events (participants affected / at risk) | 117/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous Rituximab (N=140)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 10
Atrial fibrillation (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Enterobacter bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pneumonia pneumococcal (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 4
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous Rituximab (N=140)
Anaemia (Blood and lymphatic system disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 24
Abdominal pain (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 22
Dyspepsia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 31
Injection site erythema (General disorders) | 12
Pain (General disorders) | 9
Pyrexia (General disorders) | 14
Respiratory tract infection (Infections and infestations) | 23
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 11
Viral upper respiratory tract infection (Infections and infestations) | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 15
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2013-05-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT01987505/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT01987505/SAP_001.pdf